CLINICAL TRIAL: NCT06076434
Title: The Effect on Bruising and Pain of Different Durations of Pressure Application Following Subcutaneous Heparin Injection to the Upper Arm
Brief Title: Low-Molecular-Weight Heparin Injection in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Canan Kas, PhD, MSc, RN, Assistant Professor, Kastamonu University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-KEAK-102
Record Dates: First submitted 2023-06-06; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Stroke
Keywords: Anticoagulants; Injection; Nursing
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Effect of 10 second Pressure Times on Bruising and Pain (Experimental): The patients were randomized according to age and gender and included in the groups.
  Patients were injected with heparin subcutaneously in the upper arm by the clinic nurse in accordance with the procedure of the clinic. The area was cleaned with alcohol and after the alcohol was dried, 0.6 ml of subcutaneous heparin was injected with a 27 gauge needle at a 90° angle to the tissue. The heparin was injected in approximately 10 seconds without aspirating the syringe. After injection, the area was pressurized with dry cotton wool for the specified time. After the injection, pressure was applied to the area with dry cotton for specified periods. Pain level was determined at the time of injection. Using an acetate pen, a circle of approximately 5 cm was marked around the needle insertion site and the bruising level was measured and recorded 48 hours later using a transparent film.
  Interventions: Other: The Effect of Different Pressure Periods on Bruising and Pain After Subcutaneous Heparin Injection Applied to the Upper Arm Region
- Effect of 35 second Pressure Times on Bruising and Pain (Experimental): The patients were randomized according to age and gender and included in the groups.
  Patients were injected with heparin subcutaneously in the upper arm by the clinic nurse in accordance with the procedure of the clinic. The area was cleaned with alcohol and after the alcohol was dried, 0.6 ml of subcutaneous heparin was injected with a 27 gauge needle at a 90° angle to the tissue. The heparin was injected in approximately 10 seconds without aspirating the syringe. After injection, the area was pressurized with dry cotton wool for the specified time. After the injection, pressure was applied to the area with dry cotton for specified periods. Pain level was determined at the time of injection. Using an acetate pen, a circle of approximately 5 cm was marked around the needle insertion site and the bruising level was measured and recorded 48 hours later using a transparent film.
  Interventions: Other: The Effect of Different Pressure Periods on Bruising and Pain After Subcutaneous Heparin Injection Applied to the Upper Arm Region
- Effect of 60 second Pressure Times on Bruising and Pain (Experimental): The patients were randomized according to age and gender and included in the groups.
  Patients were injected with heparin subcutaneously in the upper arm by the clinic nurse in accordance with the procedure of the clinic. The area was cleaned with alcohol and after the alcohol was dried, 0.6 ml of subcutaneous heparin was injected with a 27 gauge needle at a 90° angle to the tissue. The heparin was injected in approximately 10 seconds without aspirating the syringe. After injection, the area was pressurized with dry cotton wool for the specified time. After the injection, pressure was applied to the area with dry cotton for specified periods. Pain level was determined at the time of injection. Using an acetate pen, a circle of approximately 5 cm was marked around the needle insertion site and the bruising level was measured and recorded 48 hours later using a transparent film.
  Interventions: Other: The Effect of Different Pressure Periods on Bruising and Pain After Subcutaneous Heparin Injection Applied to the Upper Arm Region

INTERVENTIONS:
Other: The Effect of Different Pressure Periods on Bruising and Pain After Subcutaneous Heparin Injection Applied to the Upper Arm Region — The injection site on the upper arm of each patient was cleaned with alcohol and after the alcohol was dried, 0.6 ml of subcutaneous heparin was injected into the tissue at a 90° angle with a 27 gauge needle. The heparin was injected in approximately 10 seconds without aspirating the syringe. After the injection, pressure was applied to the area with dry cotton for specified periods (10 second, 35 second and 60 second).

SUMMARY:
Bruising as a result of heparin injection increases patients' anxiety, decreases their confidence in the effectiveness of nurses and causes them to refuse the injection. This undesirable effect can be reduced by using appropriate technique and taking a few simple precautions. In the systematic review conducted by İnangil and Şendir (2017) to systematically review the studies on the prevention of ecchymosis, hematoma and pain associated with subcutaneous heparin injection; it was determined that the number of studies investigating other techniques (pressure, site selection, etc.) was insufficient, with the highest number of studies on injection time and cold application. As a result of the research, it was recommended that local pressure should be applied to the area after injection, and the abdominal region should be preferred especially in patients who are sensitive to pain, since pain intensity is higher in the thigh and arm region. Due to the lack of literature, there is no consensus regarding the duration of compression to reduce bruising and pain after LMWH application. Based on these, this study was planned to compare the pressure applied to the injection point for 10, 35 and 60 seconds after injection in terms of pain, bruising and development of ecchymosis and hematoma at the injection sites in patients using subcutaneous heparin in the upper arm.

DETAILED DESCRIPTION:
Anticoagulants are medicines that prevent blood from clotting as quickly or effectively as normal. Can be administered IV or subcutaneously. The main complications of heparin therapy are bleeding, thrombocytopenia and osteoporosis. Anticoagulants are classified as Vitamin K antagonist (VKA) (oral), Unfractionated heparin (UFH) (IV or subcutaneous), LMWHD (subcutaneous), Heparinoids (IV or subcutaneous), Fondaparinux (Subcutaneous), Oral factor Xa inhibitors, Parenteral direct thrombin inhibitors and Oral direct thrombin inhibitors. Subcutaneous administration of low-molecular-weight heparin (LMWH) may cause complications such as hematoma, bruising and pain at different injection sites. It is a goal of the nurse to reduce discomfort, anxiety, worry, refusal of treatment and lack of trust in the nurse due to bruising on the skin. Several studies have been conducted to investigate whether bruising and pain depend on injection sites; however, the results are conflicting and no clear and consistent conclusion has been reached. Subcutaneous heparin injection is a common nursing clinical intervention. Nurses often inject heparin subcutaneously and this action often causes some complications such as bruising, hematoma, pain and induration at the injection site. Bruising as a result of heparin injection increases patients' anxiety, decreases their confidence in the effectiveness of nurses and causes them to refuse the injection. This undesirable effect can be reduced by using appropriate technique and taking a few simple precautions. In the systematic review conducted by İnangil and Şendir (2017) to systematically review the studies on the prevention of ecchymosis, hematoma and pain associated with subcutaneous heparin injection; it was determined that the number of studies investigating other techniques (pressure, site selection, etc.) was insufficient, with the highest number of studies on injection time and cold application. As a result of the research, it was recommended that local pressure should be applied to the area after injection, and the abdominal region should be preferred especially in patients who are sensitive to pain, since pain intensity is higher in the thigh and arm region. Due to the lack of literature, there is no consensus regarding the duration of compression to reduce bruising and pain after LMWH application. Based on these, this study was planned to compare the pressure applied to the injection point for 10, 35 and 60 seconds after injection in terms of pain, bruising and development of ecchymosis and hematoma at the injection sites in patients using subcutaneous heparin in the upper arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Hospitalized in the neurology clinic
* Who were administered at least once a day LMWH via subcutaneous injections in the arm
* Who agreed to participate in the study were included in this study

Exclusion Criteria:

* Patients who refused to participate in the study
* Patients with an INR value above 1.3 (hospital reference range was taken)
* Patients taking anticoagulant drugs were included in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
The Effect of Different Pressure Periods on Bruising and Pain After Subcutaneous Heparin Injection Applied to the Upper Arm Region | 48 hours
  In this study, in patients using LMWH on the upper arm, the pressure applied to the injection point for 10, 35 and 60 seconds after the injection, and the pain at the injection site after the pressure were measured with the Visual Analog Scale. Additionally, in patients using LMWH on the upper arm, the pressure applied to the injection point for 10, 35 and 60 seconds after injection was examined for the development of bruising, ecchymosis and hematoma 48 hours later. Researchers marked an approximately 5 cm circle around the needle entry site using an acetate pen, and the level of bruising was measured and recorded 48 hours later using clear film.

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Kastamonu, Turkey (Türkiye)